CLINICAL TRIAL: NCT03765307
Title: Safety and Efficacy of the SyMap Bronchial Ablation System for Treatment of Severe Asthma: A Prospective, Multicenter, Randomized Controlled Clinical Trial (Bronchial Ablation for Treatment of Asthma (BATA) Trial)
Brief Title: Bronchial Ablation for Treatment of Asthma (BATA) Trial
Acronym: BATA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SyMap Medical (Suzhou), Ltd. (Industry)
Collaborators: JieNuo Medical(Beijing)Co.,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201801
Record Dates: First submitted 2018-12-02; First posted 2018-12-05 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Ablation; Bronchial Thermoplasty
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Patients with severe asthma are assigned to the experimental or control group at a 1:1 ratio based on a central randomized system.
Who Masked: Participant, Outcomes Assessor
Masking Description: The enrolled patients are blinded until 12 months after procedure. Physicians who perform post-procedure patient management and physicians who perform bronchial ablation/ bronchial thermoplasty procedures are blinded to each other.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SyMap Bronchial Ablation Group (Experimental): The experimental group is treated using SyMap Bronchial Radiofrequency Ablation system, including disposable bronchial radiofrequency ablation catheter (Model: BA125T) and Bronchial radiofrequency ablation instrument (Model: ELATION S3).
  Interventions: Device: SyMap Bronchial Ablation System
- Boston Scientific Bronchial Thermoplasty Group (Active Comparator): The control group is treated using Boston Scientific Alair System, including Bronchial radiofrequency ablation catheter Alair (Model: ATS2-5 ) and Bronchial radiofrequency ablation instrument (Model: ATS200)
  Interventions: Device: Boston Scientific Alair System

INTERVENTIONS:
Device: SyMap Bronchial Ablation System — The Bronchial Ablation is performed using SyMap Bronchial Ablation System in three sessions at least three weeks apart between each session: Right Lung Lobe, Left Lung Lobe, Right Up Lobe and Left Up Lobe.
  Arms: SyMap Bronchial Ablation Group
Device: Boston Scientific Alair System — The Bronchial Thermoplasty is performed using Boston Scientific Alair System in three sessions at least three weeks apart between each session: Right Lung Lobe, Left Lung Lobe, Right Up Lobe and Left Up Lobe.
  Arms: Boston Scientific Bronchial Thermoplasty Group

SUMMARY:
To evaluate the safety and efficacy of a bronchial radiofrequency ablation system (SyMap Medical (Suzhou) Ltd) in a population of subjects with severe asthma who are still symptomatic despite being managed on high-dose Inhaled Corticosteroids (ICS) and Long-Acting β2-adrenergic Agonists (LABA).

DETAILED DESCRIPTION:
This will be a prospective, multicenter, randomized, clinical study comparing the SyMap bronchial radiofrequency ablation system to the Boston Scientific Bronchial Thermoplasty System (Alair System). The study population consisted of subjects with severe asthma who are still symptomatic despite being managed on high dose ICS and LABA. Patients with severe asthma who still have symptoms, despite the standard drug maintenance recommended by the guidelines, after signing the informed consent, who meet the inclusion exclusion criteria enter the baseline period and continued to use uniform ICS and LABA, which will last at least 4 weeks. Patients with at least two days asthma symptoms during the baseline period, and meet the eligibility criteria are assigned to the experimental or control group at a 1:1 ratio based on a central randomized system. A total of 160 subjects will be enrolled, 80 in the experimental group and 80 in the control group. The experimental group is treated with SyMap radiofrequency ablation system, and the control group is treated with the same procedure using Boston Scientific Bronchial Thermoplasty Aliar System. For subjects in the experimental group and the control group, follow-up by telephone call will be performed at 1, 2, 7 days after each procedure and at 1, 2, 4, 5, 7, 8, 9, 10, 11, 15, 18, 21, 27, 30, 33, 39, 42, 45, 51, 54, and 57 months after the third procedure, and outpatient follow-up will be performed at 6 weeks, 3, 6，12，24, 36, 48 and 60 months after the third procedure. ICS and LABA are administered within five years after the third procedure. The difference in the rate of severe asthma exacerbations per year (the number of severe asthma exacerbations per person per year), at 12 months after bronchial radiofrequency ablation, is the primary endpoint of the study, and the success rate of procedure, postoperative adverse events, and serious adverse events are safety endpoints.

This study is conducted by an independent clinical monitoring organization, a data management and statistical center to collect and statistically analyze all relevant clinical and laboratory data.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult between the ages of 18 to 65 years;
* Diagnosed with asthma who required regular asthma maintenance medication in the past 6 months as follows:

ICS ≥1000 μg/day beclomethasone or equivalent and LABA ≥1000μg /day salmeterol or equivalent.

Other medications were allowed, including leukotriene modifiers, and Oral Corticosteroids (OCS) ≤ 10mg/day.

* At least two days of asthma symptoms during 4-weeks of the baseline period.
* Pre-bronchodilator Forced Expiratory Volume in one second (FEV1) of greater than or equal to 45% of predicted.
* Non-smoker (less than 10 pack per year) last for 1 year or greater.
* Baseline AQLQ Score less than or equal to 6.25
* Willingness and ability to comply with the outpatient follow-up.

Exclusion Criteria:

* Pre-bronchodilator Forced Expiratory Volume in one second (FEV1) of less than 45% of predicted.
* 3 or more hospitalizations for exacerbations of asthma in the past 12 months;
* More than 3 lower respiratory tract infections requiring antibiotics in the past 12 months
* More than 4 of oral steroid use for exacerbations of asthma in the past 12 months
* Chronic sinusitis
* Uncontrolled gastroesophageal reflux disease, defined as a significant increase in treatment over the past 6 weeks
* Sensitivity to medications required to perform bronchoscopy (such as lidocaine and benzodiazepines)
* Use of an implantable electrical stimulation device, such as a pacemaker, a cardiac defibrillator or a deep nerve or deep brain stimulator;
* Severe emphysema caused by chronic obstructive pulmonary disease (COPD).
* Use of systemic immunosuppressants, beta adrenergic blockers, or anticoagulants.
* History of fatal asthma.
* Uncontrolled obstructive sleep apnea
* Intubation or admission to the ICU for asthma exacerbations within 2 years prior to treatment
* Hemorrhagic or malignant tumors or Coagulopathy.
* Lower bronchial stenosis or distal complete atelectasis or other severe bronchial and pulmonary lesions, as Thoracic spiral CT showed
* Poor compliance judged by the investigator, or other medical conditions that are not suitable for the study
* Related contraindications for bronchoscopy
* Pregnant, lactating women, or patients with a birth plan in the next year
* Previously undergone bronchial thermoplasty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of severe asthma exacerbations per year (the number of severe asthma exacerbations per person per year) | 12 months
  Definition of severe asthma exacerbations:
  1. Patients who do not receive oral corticosteroids maintenance, systemic corticosteroids (tablets, suspensions or injections) need to be used, or ICS doses doubled, due to increased asthma symptoms.
  2. Patients who have been treated with oral corticosteroids maintenance daily or every other day, the daily dose of systemic corticosteroids needs to be increased, due to increased asthma symptoms;
  Note: Severe asthma exacerbations of the above described two conditions, after treatment with corticosteroids, stabilized for 1 week or more, then recurring asthma symptoms will be counted as a single severe asthma exacerbations.

SECONDARY OUTCOMES:
Change in Integrated Asthma Quality of Life Questionnaire (Integrated AQLQ) Score from baseline | 3, 6, 12, 24, 36, 48 and 60 months
  Asthma Quality of Life Questionnaire consists of 32 items covering asthma-related symptoms and limitations during the 2 weeks preceding administration of the questionnaire, the responses are scored on a scale of 1 to 7, with higher numbers indicating a better quality of life. Integrated AQLQ is the average of the 6-, 9-, and 12- month scores.The proportion of subjects within each group that achieved an AQLQ score change of 0.5 or greater is analyzed.
Asthma Quality of Life Questionnaire Score (AQLQ) | 6 weeks, 3, 6, 12, 24, 36, 48 and 60months
  Asthma Quality of Life Questionnaire consists of 32 items covering asthma-related symptoms and limitations during the 2 weeks preceding administration of the questionnaire, the responses are scored on a scale of 1 to 7, with higher numbers indicating a better quality of life.
Modified Asthma Control Questionnaire (ACQ-6) Score | 6 weeks, 3, 6, 12, 24, 36, 48 and 60months
  Modified Asthma Control Questionnaire (ACQ-6) Consists of six questions (1 for bronchodilator use and 5 for asthma symptoms). The scores range from 0 (full control) to 6 (seriously uncontrolled). The ACQ-6 average score is the mean of the patient score. The average score ≤ 0.75 indicates that the asthma control is good, 0.75 ~ ≤ 1.5 prompts partial control, > 1.5 prompts poor control. The proportion of subjects within each group that achieved an AQLQ score change of 0.5 or greater was analyzed.
Percent of Symptom-Free Days | 12 months
Numbers of severe asthma exacerbations | 6 weeks, 12, 24, 36, 48 and 60 months
Forced Expiratory Volume in one second (FEV1) | 6 weeks, 12, 24, 36, 48 and 60months
Peak expiratory flow (PEF) | 6 weeks, 12 , 24, 36, 48 and 60 months
Rate of severe asthma exacerbations per year | 24, 36, 48 and 60 months
  the number of severe asthma exacerbations per person per year

OTHER OUTCOMES:
Emergency Room Visits days | 12, 24, 36, 48 and 60 months
Hospitalization days | 12, 24, 36, 48 and 60 months
Absence of work/school due to asthma symptoms, or days affecting daily actives | 12 months
Successful rate of procedure | During the procedure
  defned by whether the catheter can be engaged in the correct position in the bronchus to successfully complete the bronchial radiofrequency ablation
Safety of the procedure | During the procedure
  related adverse events and complications during the procedure
Adverse events (AEs), serious adverse events (SAEs) after procedure | 1, 2 days, and 7 days after procedure
Rate of Adverse events (AEs), serious adverse events (SAEs) | 6 weeks, 3, 6, 12, 24, 36, 48 and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue LI, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (15):
- China (15):
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - University of Chinese Academy of Sciences Shenzhen Hospital, Shenzhen, Guangdong
  - Hebei Chest Hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Affiliated Hospital Of Qiqihar Medical University, Qiqihar, Heilongjiang
  - The First Affilated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Northern Theater Command General Hospital, Shenyang, Liaoning
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Second Affiliated Hospital of Air Force Medical University, Xi’an, Shanxi
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
Our decision on whether to share the individual participant data depends on the opinions of the regulatory authorities in China, but so far the regulatory agencies have no clear instructions yet, thus we cannot make a decision at present.